CLINICAL TRIAL: NCT02402972
Title: A Multi-center Randomized Controlled Trial: Intraportal Chemotherapy Combined With Adjuvant Chemotherapy (mFOLFOX6) for Stage II and III Colon Cancer
Brief Title: A Multi-center Randomized Controlled Trial of Intraportal Chemotherapy Combined With Adjuvant Chemotherapy (mFOLFOX6) for Stage II and III Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu jianmin (Other)
Collaborators: Zhejiang University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Deputy director of the colorectal cancer center, Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IICCAC; 82345432 (Other Grant/Funding Number: Shanghai key research projects)
Record Dates: First submitted 2015-03-20; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Cancer; Metastasis
Keywords: adjuvant chemotherapy; intraportal chemotherapy; prevention
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Floxuridine; Leucovorin

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- IPC plus AC (Experimental): patients treated with intraoperative intraportal chemotherapy (IPC) plus adjuvant chemotherapy (AC; mFOLFOX6).; IPC: During the operation, one dose of fluorodeoxyuridine (FUDR) 1000 mg and oxaliplatin 100 mg were administered as a bolus into the regional vein within 5 minutes just before ligation.
  AC: All patients received mFOLFOX6 adjuvant chemotherapy, consisting of a 2-h infusion of 85 mg/m2 oxaliplatin given simultaneously with a 2-h infusion of 400 mg/m2 LV, followed by a bolus of 400 mg/m2 5-FU, and then a continuous infusion of 2000 mg/m2 5-FU given on 2 consecutive days by intravenous pumping every 14 days for 12 cycles.[1] Adverse events were categorized according to National Cancer Institute Common Toxicity Criteria, version 3.0.
  Interventions: Drug: FUDR +oxaliplatin; Drug: oxaliplatin+Leucovorin+5-FU
- AC (Active Comparator): patients treated with adjuvant chemotherapy (AC; mFOLFOX6) alone after surgery; Adjuvant chemotherapy (AC): All patients received mFOLFOX6 adjuvant chemotherapy, consisting of a 2-h infusion of 85 mg/m2 oxaliplatin given simultaneously with a 2-h infusion of 400 mg/m2 LV, followed by a bolus of 400 mg/m2 5-FU, and then a continuous infusion of 2000 mg/m2 5-FU given on 2 consecutive days by intravenous pumping every 14 days for 12 cycles.[1] Adverse events were categorized according to National Cancer Institute Common Toxicity Criteria, version 3.0.
  Interventions: Drug: oxaliplatin+Leucovorin+5-FU

INTERVENTIONS:
Drug: FUDR +oxaliplatin — IPC: one dose of fluorodeoxyuridine (FUDR) 1000 mg and oxaliplatin 100 mg were administered as a bolus into the regional vein
  Other Names: fluorodeoxyuridine (FUDR)
  Arms: IPC plus AC
Drug: oxaliplatin+Leucovorin+5-FU — Adjuvant chemotherapy (AC): All patients received mFOLFOX6 adjuvant chemotherapy: oxaliplatin+Leucovorin+5-FU
  Other Names: Leucovorin (LV)

SUMMARY:
To investigate whether intraoperative intraportal chemotherapy combined with adjuvant chemotherapy as treatment could improve disease-free survival (DFS) in patients with curative colorectal cancer resection compared with adjuvant chemotherapy alone.

This is a prospective, blind (doctors who done outcome measures were masked), multi-center, 2-arm randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Primary tumor has undergone histologically confirmed colon adenocarcinoma; Colon cancer was defined by the presence of the inferior pole of the tumor above the peritoneal reflection (at least 15 cm from the anal margin).
3. Together with clinical or radiological evidence of Stage II (T3-4, N0, M0) or Stage III (T1-4, N1-2, M0) disease (according to the 2007 revision of the International Union Against Cancer TNM staging system)
4. Performance status (ECOG) 0~1
5. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; Hb ≥9g/dl (within 1 week prior to randomization)
6. Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either AST or ALT) ≤ 5 x ULN(within 1 week prior to randomization);
7. Written informed consent for participation in the trial.

Exclusion Criteria:

1. Previous exposure to prior cancer therapy (chemotherapy, radiotherapy or intervention therapy) for colon cancer.
2. Patients with known hypersensitivity reactions to any of the components of the study treatments.
3. Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
4. Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
5. Known drug abuse/ alcohol abuse
6. Legal incapacity or limited legal capacity
7. Pre-existing peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | up to 5 year
  DFS was defined as from the date of randomization to the date of tumor recurrence or death from any cause.

SECONDARY OUTCOMES:
overall survival | 3 year and 5 year
  OS was measured from the date of randomization to the date of death from any cause.
metastasis-free survival | 3 year and 5 year
  MFS was defined as the time from randomization to metastasis if metastasis was the first event.
adverse events of Chemotherapy and IPC | 6 months
  toxicity (using NCI CTC 3.0) compared with mFOLFOX6 alone.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, MD, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China